CLINICAL TRIAL: NCT01539902
Title: A Randomized, Double Blind, Parallel Group, Placebo Controlled Research of Human Umbilical Cord Derived Mesenchymal Stem Cell for the Treatment of Lupus Nephritis
Brief Title: Phase 2 Study of Human Umbilical Cord Derived Mesenchymal Stem Cell for the Treatment of Lupus Nephritis
Acronym: hUC-MSC-SLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CytoMed & Beike (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT 11-03
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Lupus Nephritis
Keywords: MSC for the treatment of Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Umbilical Cord derived MSCs (Experimental)
  Interventions: Biological: Human Umbilical Cord derived MSCs
- Cyclophosphamide (Placebo Comparator)
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Human Umbilical Cord derived MSCs — Human Umbilical Cord derived MSCs treatment for lupus nephritis via infusion
  Other Names: Allogeneic stem cells derived from umbilical cord
  Arms: Human Umbilical Cord derived MSCs
Drug: Cyclophosphamide — Cyclophosphamide based immunosuppressive agent for treatment for lupus nephritis
  Other Names: Immunosupressive agent
  Arms: Cyclophosphamide

SUMMARY:
The efficacy measure of hUC-MSC in the treatment of proliferative lupus nephritis on remission of lupus nephritis (combined partial and complete remission) in terms of stabilization and improvement in renal function.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Male or non-pregnant females age 16 to 65 years inclusive.
2. Written informed consent obtained from patient or parents/guardian.
3. Patients with SLE fulfilling American Rheumatism Association criteria and SLEDAI score>8 or BILAG score A/B.
4. Patients with newly diagnosed World Health Organization (WHO) Class III or IV Lupus Nephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant females age 16 to 65 years inclusive.
2. Written informed consent obtained from patient or parents/guardian.
3. Patients with SLE fulfilling American Rheumatism Association criteria and SLEDAI score>8 or BILAG score A/B.
4. Patients with newly diagnosed World Health Organization (WHO) Class III or IV Lupus Nephritis

Exclusion Criteria:

Patients with any of the following are not eligible for enrollment into the study:

1. Pregnant or nursing woman or women of childbearing potential except if post-menopausal, surgically sterile or using accepted method(s) of birth control or having negative pregnancy test.
2. Participation in any research in which the patient received an investigational product within 30 days preceding the screening phase of this study.
3. Those persons directly involved in the conduct of the study.
4. Serum creatinine more than 250 µmol/L.
5. White blood cell (WBC) count of less than 3.5 X 109/L.
6. Active peptic ulcer disease.
7. Active systemic infection.
8. History of alcohol or substance abuse.
9. History of malignancy within previous 5 years.
10. Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of this study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy and Safety | 6 months
  The efficacy measure is remission of nephritis (combined partial and complete remission) at 6 months defined as
  * Stabilization or improvement in renal function and
  * Urinary RBC of less than 10 per HPF and
  * Reduction of proteinuria to less than 3 g/day if baseline proteinuria was more than 3 g/day and at least a 50% reduction in proteinuria, or to less than 1 g/day if the baseline proteinuria was in the subnephrotic range.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital & SLE Research Centre, Kunming Medical University, Kunming China, Kunming, Yunan, China

REFERENCES:
- [Derived] Deng D, Zhang P, Guo Y, Lim TO. A randomised double-blind, placebo-controlled trial of allogeneic umbilical cord-derived mesenchymal stem cell for lupus nephritis. Ann Rheum Dis. 2017 Aug;76(8):1436-1439. doi: 10.1136/annrheumdis-2017-211073. Epub 2017 May 6. PMID 28478399